CLINICAL TRIAL: NCT03087552
Title: Safety and Feasibility of Transradial Mini-invasive Balloon Aortic Valvuloplasty
Brief Title: Mini-invasive Balloon Aortic Valvuloplasty
Acronym: SOFTLY-II
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, University Hospital of Ferrara
Other Study IDs: 18072011
Record Dates: First submitted 2017-03-11; First posted 2017-03-22 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transradial balloon aortic valvuloplasty: Consecutive patients with severe aortic stenosis and receiving as first attempt balloon aortic valvuloplasty by transradial access.
  Interventions: Procedure: Transradial balloon aortic valvuloplasty

INTERVENTIONS:
Procedure: Transradial balloon aortic valvuloplasty — Mini-invasive balloon aortic valvuloplasty consisting in transradial access
Procedure: Transradial balloon aortic valvuloplasty — Rapid pacing using the 0.035-in. retrograde left ventricular support wire

SUMMARY:
The spreading of transcatheter aortic valve implantation has paradoxically increased the spectrum of indications for balloon aortic valvuloplasty. Balloon aortic valvuloplasty is currently used as destination therapy for patients excluded from transcatheter aortic valve implantation, as bridge to transcatheter aortic valve implantation or to surgical aortic valve replacement, or as a stratification tool for selected high-risk patients who cannot be immediate candidates for transcatheter aortic valve implantation. Moreover, it has been recently showed that transcatheter aortic valve implantation without balloon aortic valvuloplasty is encumbered by an increased risk of cerebral embolization. However, balloon aortic valvuloplasty has a complication rate comparable to transcatheter aortic valve implantation, mainly related to access site or temporary pacemaker implantation. Thus, a transradial mini-invasive approach with rapid pacing through the 0,035 inch left ventricular support wire could be extremely appealing.

DETAILED DESCRIPTION:
Consecutive patients with severe aortic stenosis with indication to aortic balloon valvuloplasty will be enrolled. An ad hoc informed consent for the procedure will be obtained from all patients.

This is a prospective observational study. The Investigators will include patients where aortic ballloon valvuloplasty is attempted by radial access and without temporary pacemaker implantation. The aim is to register and monitor the effectiveness and safety of this approach. Details regarding management of radial access and pacing with 0.035 wire can be found in the references reported below. The primary endpoint will be the 30-day occurence of minor and major vascular complications according VARC 2 classification. The safety endpoint will be the absence of intra- or periprocedural major complications in transradial balloon aortic valvuloplasty, namely balloon entrapment or compartment syndrome requiring surgical intervention.

The feasibility endpoint will be a procedural success rate ≥90%. The efficacy endpoint will be a reduction of the mean invasive gradient >30%. At baseline, Handgrip strength test will be performed and angiography of the instrumented arm will be performed at the beginning and at the end of the procedure. All patients will be prospectively followed-up for at least 30 days and all adverse events will be recorded. All patients will be assessed also for frailty according the clinical frailty scale (CFS). During the 30-day follow-up visit two independent blinded operators will evaluate radial artery patency by ultrasonography and perform handgrip strength test in in both arms in all patients.

ELIGIBILITY:
Inclusion Criteria:

* severe symptomatic aortic stenosis requiring balloon aortic valvuloplasty

Exclusion Criteria:

* cardiogenic shock
* bilateral absence of radial pulse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe aortic stenosis with indication to balloon aortic valvuloplasty
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2017-03-11 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Vascular complications | 1 month
  Cumulative occurrence of major and minor bleeding complications according the VARC-2 classification

SECONDARY OUTCOMES:
Transradial balloon aortic valvuloplasty major complications | 1 month
  Balloon entrapment, compartment syndrome requiring surgical intervention
Adverse events | 1 month
  Cumulative occurrence of death, stroke, coronary occlusion, coronary dissection, moderate-severe aortic regurgitation, severe hypotension requiring intervention, pericardiocentesis, definitive pace-maker implantation
Major vascular complications | 1 month
  Cumulative occurrence of major bleeding complications according the VARC-2
Minor vascular complications | 1 month
  Cumulative occurrence of minor bleeding complications according the VARC-2
Radial artery occlusion | 1 month
  Cumulative occurrence of radial artery occlusion
Radial artery occlusion | 24 hours
  Cumulative occurrence of radial artery occlusion

OTHER OUTCOMES:
Frailty assessment | 1 month
  Improvement from baseline to 1 month of the Clinical Frailty Scale. The Clinical Frailty Scale (CFS) ranges from 1 to 9, with higher values suggestive for poor prognosis
Physical performance assessment | 1 month
  Improvement from baseline to 1 month of grip strength
Essential Frailty Toolset | 1 month
  Improvement from baseline to 1 month of the value of the Essential Frailty Toolset scale. The Essential Frailty Toolset (EFT) ranges from 0 to 5, with higher values suggestive for poor prognosis

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (17):
  - University Hospital of Ferrara, Cona, Ferrara
  - Pia Fondazione Panico, Tricase, Lecce
  - Ospedale Bassini, Cinisello Balsamo, Milano
  - AOU San Luigi Gonzaga, Orbassano, Torino
  - Ospedale di Conegliano, Conegliano, Treviso
  - AOU di Ancona, Ancona
  - AOU di Bologna, Bologna
  - Ospedale Morgagni Pierantoni, Forlì
  - Ospedale Misericordia, Grosseto
  - Ospedale Vito Fazzi, Lecce
  - Ospedale Civile Santo Spirito, Pescara
  - Ospedale Santa Maria delle Croci, Ravenna
  - Ospedale degli Infermi, Rimini
  - Ospedale San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Ospedale di Sassari, Sassari
  - ASL di Teramo, Teramo
  - Ospedale degli Infermi di Rivoli, Torino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tumscitz C, Pirani L, Tebaldi M, Campo G, Biscaglia S. Seven french radial artery access for PCI: a prospective single-center experience. Int J Cardiol. 2014 Oct 20;176(3):1074-5. doi: 10.1016/j.ijcard.2014.07.134. Epub 2014 Aug 2. No abstract available. PMID 25127334
- [Background] Hilling-Smith R, Cockburn J, Dooley M, Parker J, Newton A, Hill A, Trivedi U, de Belder A, Hildick-Smith D. Rapid pacing using the 0.035-in. Retrograde left ventricular support wire in 208 cases of transcatheter aortic valve implantation and balloon aortic valvuloplasty. Catheter Cardiovasc Interv. 2017 Mar 1;89(4):783-786. doi: 10.1002/ccd.26720. Epub 2016 Oct 11. PMID 27726292
- [Derived] Tumscitz C, Di Cesare A, Balducelli M, Piva T, Santarelli A, Saia F, Tarantino F, Preti G, Picchi A, Rolfo C, Attisano T, Colonna G, De Iaco G, Parodi G, Di Marco M, Cerrato E, Pierini S, Fileti L, Cavazza C, Dall'Ara G, Govoni B, Mantovani G, Serenelli M, Penzo C, Tebaldi M, Campo G, Biscaglia S. Safety, efficacy and impact on frailty of mini-invasive radial balloon aortic valvuloplasty. Heart. 2021 Jun;107(11):874-880. doi: 10.1136/heartjnl-2020-318548. Epub 2021 Feb 24. PMID 33627400